CLINICAL TRIAL: NCT01367860
Title: Comparison of Percutaneous Diskectomy SpineJet x Open Microdiscectomy for Treatment of Lumbar Radiculopathy in Contained Disc Herniation: Randomized Clinical Trial
Brief Title: Percutaneous Diskectomy SpineJet x Open Microdiskectomy in Treatment of Lumbar Radiculopathy
Acronym: PDOP_TLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alexandre F. Cristante, PhD., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SpJet2011; IOT (Other: iot 803 [institutional research committee])
Record Dates: First submitted 2011-05-31; First posted 2011-06-07 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Radiculopathy; Herniated Disk
Keywords: spine surgery; low back pain; herniated disk
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMicro (Active Comparator): This group will be formed by randomization, which gets out surgery to open microdiscectomy
  Interventions: Procedure: Open microdiscectomy
- SJet (Experimental): This group will be formed by randomization, and receive the discectomy procedure addressed by the technique of Percutaneous Diskectomy SpineJet
  Interventions: Procedure: Percutaneous Diskectomy SpineJet

INTERVENTIONS:
Procedure: Open microdiscectomy — The open microdiscectomy, will be performed under general anesthesia in the prone position with horizontal. The level of the spine indicated for surgical treatment will be identified with the aid of fluoroscopy. An incision is made about the dorsal disc level involved with dissection of the paravertebral muscles on the side of disc herniation. After laminectomy and resection of part of the yellow ligament, partial discectomy is done under direct vision.
  Arms: OMicro
Procedure: Percutaneous Diskectomy SpineJet — Percutaneous Diskectomy SpineJet be performed under local anesthesia, in which a needle is placed via percutaneous posterolateral extra-pedicular, below the neural foramen in the center of the disc, using the traditional approach for discography. The researcher will confirm the proper placement of the needle in front and side incidences on the fluoroscopy.
  Arms: SJet

SUMMARY:
Approximately 300,000 patients undergo open surgical procedures to treat symptoms caused by disc herniation.

Among the various surgical techniques practiced the percutaneous discectomy occupies its space since the first description of the technique by Hijikata, 1975. Throughout, many techniques have been described. Studies indicate that the treatment was successful for pain and disability resulting from herniated disc associated with radiculopathy small.

However, some methods remove very small amounts of tissue with little change in volume of the disc. Thus, studies on the cadaver with Percutaneous Diskectomy by SpineJet ® showed more macroscopic changes of the disc with a predictable amount of removal and significant disc material.

The Percutaneous Diskectomy by SpineJet ® is a new technique of percutaneous diskectomy which creates a suction effect in tissues adjacent to the exit point of the fluid and the opening point of the collector. However, no studies have examined the effect of the Percutaneous Diskectomy by SpineJet ® in humans about the disk size after treatment or measures of disc degeneration by imaging methods or how these characteristics might correlate with clinical outcomes.

Thus, the study will compare outcomes of patients with contained or extruded disc herniation, with complaints of radiculopathy, concordant with the imaging findings. With treatment by surgical technique or the traditional by SpineJet ®, in order to determine whether percutaneous discectomy with SpineJet ® will produce results comparable to open microdiskectomy.

ELIGIBILITY:
Inclusion Criteria:

* single disc herniation, posterolateral, at any lumbar level, with a size of up to 1 / 3 of the spinal canal sagittal diameter, with radicular pain correlated with findings at MRI
* Failure of nonoperative treatment with at least one anti-inflammatory medication and at least two weeks of physical therapy within a period of 6 months
* acceptance of completion of informed consent

Exclusion Criteria:

* Force <4 / 5 in a muscle group in the lower limb
* Herniated Disc extrusa large (> 1 / 3 of the sagittal canal diameter) or sequestered herniation
* moderate to grade stenosis of the central canal, lateral recess or foramen
* Surgery in the previous level involved
* Herniated disc at another level in the affected side
* Loss of disc height significantly (> 60%) compared with the adjacent higher level
* Infection at the insertion of the device
* Pregnancy
* Any illness or medications that contraindicate surgical treatment

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Orthopedics and Traumatology of the USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Hijikata S, Yamagishi M, Nakayama T, Oomori K. Percutaneous nucleotomy: a new treatment method for lumbar disk herniation. J Toden Hosp 1976, 6:6-13
- [Background] Choy DS, Hellinger J, Tassi GP, Hellinger S. Percutaneous laser disc decompression. Photomed Laser Surg. 2007 Feb;25(1):60. doi: 10.1089/pho.2006.9999. No abstract available. PMID 17352640
- [Background] Davis GW, Onik G. Clinical experience with automated percutaneous lumbar discectomy. Clin Orthop Relat Res. 1989 Jan;(238):98-103. PMID 2521319
- [Background] Mochida J, Toh E, Nomura T, Nishimura K. The risks and benefits of percutaneous nucleotomy for lumbar disc herniation. A 10-year longitudinal study. J Bone Joint Surg Br. 2001 May;83(4):501-5. doi: 10.1302/0301-620x.83b4.11508. PMID 11380118
- [Background] Choy DS. Percutaneous laser disc decompression (PLDD): 352 cases with an 8 1/2-year follow-up. J Clin Laser Med Surg. 1995 Feb;13(1):17-21. doi: 10.1089/clm.1995.13.17. PMID 10150569
- [Background] Wang JC, Shapiro MS, Hatch JD, Knight J, Dorey FJ, Delamarter RB. The outcome of lumbar discectomy in elite athletes. Spine (Phila Pa 1976). 1999 Mar 15;24(6):570-3. doi: 10.1097/00007632-199903150-00014. PMID 10101821
- [Background] Pauza KJ, Howell S, Dreyfuss P, Peloza JH, Dawson K, Bogduk N. A randomized, placebo-controlled trial of intradiscal electrothermal therapy for the treatment of discogenic low back pain. Spine J. 2004 Jan-Feb;4(1):27-35. doi: 10.1016/j.spinee.2003.07.001. PMID 14749191
- [Background] Casey KF, Chang MK, O'Brien ED, Yuan HA, McCullen GM, Schaffer J, Kambin P. Arthroscopic microdiscectomy: comparison of preoperative and postoperative imaging studies. Arthroscopy. 1997 Aug;13(4):438-45. doi: 10.1016/s0749-8063(97)90121-3. PMID 9276049
- [Background] Delamarter RB, Howard MW, Goldstein T, Deutsch AL, Mink JH, Dawson EG. Percutaneous lumbar discectomy. Preoperative and postoperative magnetic resonance imaging. J Bone Joint Surg Am. 1995 Apr;77(4):578-84. doi: 10.2106/00004623-199504000-00011. PMID 7713975
- [Background] Tonami H, Yokota H, Nakagawa T, Higashi K, Okimura T, Yamamoto I, Nishijima Y. Percutaneous laser discectomy: MR findings within the first 24 hours after treatment and their relationship to clinical outcome. Clin Radiol. 1997 Dec;52(12):938-44. doi: 10.1016/s0009-9260(97)80228-0. PMID 9413969
- [Background] Krugluger J, Knahr K. Chemonucleolysis and automated percutaneous discectomy--a prospective randomized comparison. Int Orthop. 2000;24(3):167-9. doi: 10.1007/s002640000139. PMID 10990391
- [Background] Vigatto R, Alexandre NM, Correa Filho HR. Development of a Brazilian Portuguese version of the Oswestry Disability Index: cross-cultural adaptation, reliability, and validity. Spine (Phila Pa 1976). 2007 Feb 15;32(4):481-6. doi: 10.1097/01.brs.0000255075.11496.47. PMID 17304141
- [Background] Dullerud R, Nakstad PH. Side effects and complications of automated percutaneous lumbar nucleotomy. Neuroradiology. 1997 Apr;39(4):282-5. doi: 10.1007/s002340050410. PMID 9144678
- [Background] Wittenberg RH, Oppel S, Rubenthaler FA, Steffen R. Five-year results from chemonucleolysis with chymopapain or collagenase: a prospective randomized study. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1835-41. doi: 10.1097/00007632-200109010-00002. PMID 11568690
- [Result] Slotman GJ, Stein SC. Laminectomy compared with laparoscopic diskectomy and outpatient laparoscopic diskectomy for herniated L5-S1 intervertebral disks. J Laparoendosc Adv Surg Tech A. 1998 Oct;8(5):261-7. doi: 10.1089/lap.1998.8.261. PMID 9820717
- [Result] Amoretti N, Huchot F, Flory P, Brunner P, Chevallier P, Bruneton JN. Percutaneous nucleotomy: preliminary communication on a decompression probe (Dekompressor) in percutaneous discectomy. Ten case reports. Clin Imaging. 2005 Mar-Apr;29(2):98-101. doi: 10.1016/j.clinimag.2004.10.024. PMID 15752964
- [Result] Matsui H, Aoki M, Kanamori M. Lateral disc herniation following percutaneous lumbar discectomy. A case report. Int Orthop. 1997;21(3):169-71. doi: 10.1007/s002640050143. PMID 9266296
- [Result] Mayer HM, Brock M. Percutaneous endoscopic discectomy: surgical technique and preliminary results compared to microsurgical discectomy. J Neurosurg. 1993 Feb;78(2):216-25. doi: 10.3171/jns.1993.78.2.0216. PMID 8267686
- [Result] Teng GJ, Jeffery RF, Guo JH, He SC, Zhu HZ, Wang XH, Wu YZ, Lu JM, Ling XL, Qian Y, Zhang YM, Zhu MJ, Guan L, He XM. Automated percutaneous lumbar discectomy: a prospective multi-institutional study. J Vasc Interv Radiol. 1997 May-Jun;8(3):457-63. doi: 10.1016/s1051-0443(97)70589-x. PMID 9152922
- [Result] Bernhardt M, Gurganious LR, Bloom DL, White AA 3rd. Magnetic resonance imaging analysis of percutaneous discectomy. A preliminary report. Spine (Phila Pa 1976). 1993 Feb;18(2):211-7. PMID 8441936
- [Derived] Cristante AF, Rocha ID, MartusMarcon R, Filho TE. Randomized clinical trial comparing lumbar percutaneous hydrodiscectomy with lumbar open microdiscectomy for the treatment of lumbar disc protrusions and herniations. Clinics (Sao Paulo). 2016 May;71(5):276-80. doi: 10.6061/clinics/2016(05)06. PMID 27276397
- [Derived] Rocha ID, Cristante AF, Marcon RM, Oliveira RP, Letaif OB, Barros Filho TE. Controlled medial branch anesthetic block in the diagnosis of chronic lumbar facet joint pain: the value of a three-month follow-up. Clinics (Sao Paulo). 2014 Aug;69(8):529-34. doi: 10.6061/clinics/2014(08)05. PMID 25141111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred to our tertiary hospital for lumbar back pain were recruited. They were included in the study if they had disc protrusion or small herniation in only one level, with magnetic resonance imaging findings compatible with symptoms, without neurological deficits, and with no resolution after six weeks of conservative treatment.
Pre-assignment Details: Exclusion criteria were: neurological changes during conservative treatment, pregnancy, clinical status not adequate for surgical procedures, non-adherence to informed consent form. After inclusion in the study, patients were evaluated for pain and function and then randomly allocated in two groups
Groups:
- OMicro: This group will be formed by randomization, which gets out surgery to open microdiscectomy
  Open microdiscectomy : The open microdiscectomy, will be performed under general anesthesia in the prone position with horizontal. The level of the spine indicated for surgical treatment will be identified with the aid of fluoroscopy. An incision is made about the dorsal disc level involved with dissection of the paravertebral muscles on the side of disc herniation. After laminectomy and resection of part of the yellow ligament, partial discectomy is done under direct vision.
- SJet: This group will be formed by randomization, and receive the discectomy procedure addressed by the technique of Percutaneous Diskectomy SpineJet
  Percutaneous Diskectomy SpineJet : Percutaneous Diskectomy SpineJet be performed under local anesthesia, in which a needle is placed via percutaneous posterolateral extra-pedicular, below the neural foramen in the center of the disc, using the traditional approach for discography. The researcher will confirm the proper placement of the needle in front and side incidences on the fluoroscopy.
Period: Overall Study
Arm/Group | OMicro | SJet
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMicro | SJet | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (9.3) | 44.9 (9.4) | 43 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 17 | 13 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40
Schooling [Number; unit: participants] — Schooling (>=8 years and <8 years)
  participants
    >=8 years | 10 | 10 | 20
    <8 years | 10 | 10 | 20
Married [Number; unit: participants]
  Yes | 18 | 13 | 31
  No | 2 | 7 | 9
Manual labor [Number; unit: participants]
  yes | 13 | 12 | 25
  no | 7 | 8 | 15
Opioid use [Number; unit: participants]
  yes | 13 | 11 | 24
  no | 7 | 9 | 16
Working currently [Number; unit: participants]
  yes | 6 | 10 | 16
  no | 14 | 10 | 24
Receiving government benefit [Number; unit: participants]
  yes | 13 | 10 | 23
  no | 7 | 10 | 17
Months away from work [Mean (Standard Deviation); unit: Months] | 4.65 (6.52) | 8.67 (14.4) | 5.8 (9.14)
Months feeling pain [Mean (Standard Deviation); unit: Months] | 16.25 (20.2) | 33.5 (47.3) | 24.87 (36.96)
VAS for lumbar pain preoperatively [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) -> minimum value=0 and maximum value=100, higher values represent a worse outcome and zero is a better outcome.
  units on a scale | 77.2 (27) | 63 (30) | 69.2 (29)
VAS for leg pain preoperatively [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) -> minimum value=0 and maximum value=100, higher values represent a worse outcome and zero is a better outcome.
  units on a scale | 84.2 (23) | 73.6 (22) | 78.9 (22)
ODI preoperatively [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index (ODI) -> The Oswestry Disability Index (ODI) is one of the principal condition-specific outcome measures used in the management of spinal disorders. The ODI is the most commonly outcome measures in patients with low back pain.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. If the FIRST statement is marked, the section score = 0, If the LAST statement is marked, it = 5.
  0 is the best outcome and 50 is the worst outcome.
  units on a scale | 33.65 (9.33) | 26.35 (6.6) | 30 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: VAS for Lumbar Pain in 3 Months
Description: Pain Score - Visual Analog Scale (VAS) -> minimum value=0 and maximum value=10, higher values represent a worse outcome and zero is a better outcome.
Time Frame: VAS for Lumbar Pain at 3 Months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 2.63 (2.9) | 4.53 (3.47)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-4.05 to 0.26], Standard Error of Mean 1.06

2. Secondary Outcome: Clinical Evaluation
Description: Will be measured dichotomously: (present or absent)
  Variables:
  Infection; residual pain; herniation recurrency
Time Frame: 6th month
Population: Infection
Measure: Number; unit: participants
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
participants
  Infection | 1 | 1
  residual pain | 3 | 4
  herniation recurrency | 2 | 1
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, Fisher Exact

3. Secondary Outcome: VAS for Lumbar - 1st Week
Description: as for outcome 1
Time Frame: 1st week from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 3.71 (2.76) | 4.1 (2.93)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-2.21 to 1.43], Standard Error of Mean 0.90

4. Secondary Outcome: VAS for Lumbar 1st Month
Description: as for outcome 1
Time Frame: 1st month from surgery
Population: intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 3.34 (2.92) | 4.06 (3.31)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-2.76 to 1.33], Standard Error of Mean 1.01

5. Secondary Outcome: VAS for Lumbar Pain - 3rd Month
Description: as for outcome 1
Time Frame: 3rd month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 2.63 (2.9) | 4.53 (3.47)

6. Secondary Outcome: VAS for Lumbar Pain - 6th Month
Description: as for outcome 1
Time Frame: 6th month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 3.5 (3.54) | 3.79 (3.34)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-2.58 to 2.01], Standard Error of Mean 1.13

7. Secondary Outcome: VAS for Lumbar Pain - 12th Month
Description: as for outcome 1
Time Frame: 12th month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 4.06 (3.54) | 3.03 (3.32)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-1.3 to 3.3], Standard Error of Mean 1.14

8. Secondary Outcome: Oswestry Disability Index (ODI) - 1st Week
Description: Oswestry Disability Index (ODI) -> The Oswestry Disability Index (ODI) is one of the principal condition-specific outcome measures used in the management of spinal disorders. The ODI is the most commonly outcome measures in patients with low back pain.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. If the FIRST statement is marked, the section score = 0, If the LAST statement is marked, it = 5.
  0 is the best outcome and 50 is the worst outcome.
Time Frame: 1st week minus baseline
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 23.25 (9.37) | 20 (8.13)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Median Difference (Final Values) = 3.2, 95% CI 2-sided [-2.36 to 8.8], Standard Error of Mean 2.77

9. Secondary Outcome: Oswestry Disability Index (ODI) - 1st Month
Description: as for outcome 8
Time Frame: 1st month from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 19.25 (10.23) | 10.78 (2.41)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Median Difference (Final Values) = 2.2, 95% CI 2-sided [-4.4 to 8.9], Standard Error of Mean 3.3

10. Primary Outcome: Oswestry Disability Index (ODI) - 3th Month
Description: as for outcome 8
Time Frame: 3th month
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 17.05 (10.9) | 16.85 (12)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-7.15 to 7.55], Standard Error of Mean 3.6

11. Secondary Outcome: Oswestry Disability Index (ODI) - 6th Month
Description: as for outcome 8
Time Frame: 6th month from surgery
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 15.37 (11.45) | 15.1 (11.37)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-7.14 to 7.67], Standard Error of Mean 3.65

12. Secondary Outcome: Oswestry Disability Index (ODI) - 12th Month
Description: as for outcome 8
Time Frame: 12th month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 11 (6.82) | 12.7 (12.2)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-8.16 to 4.76], Standard Error of Mean 3.18

13. Secondary Outcome: VAS for Leg Pain - 1st Week
Description: Pain Score for leg pain- Visual Analog Scale (VAS) -> minimum value=0 and maximum value=10, higher values represent a worse outcome and zero is a better outcome.
Time Frame: 1st week from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 4.3 (2.92) | 2.61 (2.67)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-0.12 to 3.46], Standard Error of Mean 0.88

14. Secondary Outcome: VAS for Leg Pain - 1st Month
Description: Pain Score for leg pain - Visual Analog Scale (VAS) -> minimum value=0 and maximum value=10, higher values represent a worse outcome and zero is a better outcome.
Time Frame: 1st month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 2.96 (3.4) | 2.76 (3.41)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-2 to 2.4], Standard Error of Mean 1.09

15. Secondary Outcome: VAS for Leg Pain - 3rd Month
Description: as for outcome 14
Time Frame: 3rd month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 17.05 (10.9) | 16.85 (12)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-2.55 to 1.85], Standard Error of Mean 1.08

16. Secondary Outcome: VAS for Leg Pain - 6rd Month
Description: as for outcome 14
Time Frame: 6th month from surgery
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 2.84 (3.82) | 2.88 (3.14)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-2.29 to 2.23], Standard Error of Mean 1.11

17. Secondary Outcome: VAS for Leg Pain - 12th Month
Description: pain scale - VAS for leg pain - 12th month
Time Frame: 12th month from surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMicro | SJet
Number analyzed (Participants) | 20 | 20
units on a scale | 3.37 (3.8) | 2.67 (3.3)
Statistical Analysis 1: Comparison: OMicro vs SJet; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.67 to 3.08], Standard Error of Mean 1.17

ADVERSE EVENTS:
Arm/Group | OMicro | SJet
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No